CLINICAL TRIAL: NCT07010029
Title: Coronary Sinus Reducer in Patients With Angina With no Obstructive Coronary Disease: a Prospective Single-arm Study
Brief Title: Coronary Sinus Reducer in Patients With Angina With no Obstructive Coronary Disease
Acronym: REDUCE-ANOCA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Mariusz Tomaniak, Professor, Medical University of Warsaw
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REDUCE-ANOCA
Record Dates: First submitted 2025-05-23; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Angina With No Obstructive Coronary Artery Disease; ANOCA; Coronary Sinus Reducer
Keywords: CFR; IMR; Angina; ANOCA; CSR; Coronary Sinus Reducer; Diastolic Dysfunction; Quality of Life; FFR
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Intervention Model Description: Prospective, single-arm cohort study including patients with angina with no obstructive coronary artery disease. Enrolled patients will undergo the Neovasc reducer implantation with periprocedural evaluation of coronary microcirculation (continous thermodilution) before and directly after the device implantation. All patients will be assessed with echocardiography (evaluation by external corelab) at baseline and at six months of follow-up. Patients will also undergo exercise testing (six-minute walk test) and assessment of quality of life (SF-36), as well as angina severity (Seattle Angina Questionnaire, Dedicated app and Canadian Cardiovascular Society grade).
  Patients will also undergo the prolonged two-years follow-up (long term follow-up) regarding angina severity and QoL to evaluate the persistence of the effect - those outcomes will be included in separate analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Coronary Sinus Reducer (Experimental): Patients will undergo implantation of Coronary Sinus Reducer
  Interventions: Device: Coronary Sinus Reducer

INTERVENTIONS:
Device: Coronary Sinus Reducer — Patients will undergo implantation of Coronary Sinus Reducer

SUMMARY:
Even half of patients with angina undergoing invasive coronary angiography presents without any significant epicardial stenosis. In these cases, symptoms are usually caused by coronary microvascular dysfunction (CMD), developing as a result of several potential underlying pathophysiologies. A wide range of underlying pathomechanisms makes it challenging to develop molecular-targeted pharmacological solutions; thus, direct physiology modification has been introduced as a promising concept. The coronary sinus reducer (CSR) narrows the coronary sinus, which causes symptom relief in patients with refractory angina and coronary stenosis. CSR implantation aims to increase the coronary sinus pressure, which raises venous back pressure into the myocardium. Despite several hypotheses, the exact physiological mechanisms remain not fully elucidated. Recent data from observational studies also suggest the beneficial effect of CMD on microvascular indices. To date, there are limited data regarding the efficacy of this solution in patients with angina with no obstructive coronary artery disease (ANOCA). Of note, patients with ANOCA are frequently burdened with other comorbidities, such as heart failure with preserved ejection fraction (HFpEF). HFpEF presence relates to worse prognosis and higher risk of future cardiovascular events. Previous works showed that HFpEF is significantly associated with the appearance of CMD. Due to the small variety of drugs for HFpEF, treatment targeting CMD may be a promising therapeutic target for this disease. To date, there is also no data regarding the impact of CSR implantation on function of left ventricle and echocardiographic indexes impaired in diastolic dysfunction in patients with ANOCA. Proposed study aims to evaluate the CSR as a therapeutic strategy in patients with ANOCA to improve angina, as well as quality of life and will deliver the results regarding CSR impact on diastolic function of left and right ventricle. This study will also evaluate the mechanisms standing behind the benefits of CSR use. Neovasc reducer produced by Shockwave Medical inc will be used as CSR device in this study. Proposed study may lead to the introduction of the Neovasc reducer to the guidelines for ANOCA patients. It will also provide the data on Neovasc reducer potential use as a supportive therapy in patients with HFpEF. Prospective, single-arm cohort study including patients with angina with no obstructive coronary artery disease. Enrolled patients will undergo the Neovasc reducer implantation with periprocedural evaluation of coronary microcirculation before and directly after the device implantation. All patients will be assessed with echocardiography (evaluation by external corelab) at baseline and at six months of follow-up. Patients will also undergo exercise testing (six-minute walk test) and assessment of quality of life (SF-36), as well as angina severity (Seattle Angina Questionnaire, Dedicated app and Canadian Cardiovascular Society grade).

ELIGIBILITY:
Inclusion Criteria:

* Stable angina symptoms without significant obstruction of coronary artery (defined as coronary artery stenosis diameter ≤ 50% or coronary artery stenosis diameter >50% and ≤70% with FFR>0.8), with coronary microvascular dysfunction confirmed in invasive test (defined as coronary flow reserve ≤ 2.5 or index of microvascular resistance ≥ 25)
* No future options for antianginal therapy (maximum antianginal therapy for at least three months)

Exclusion Criteria:

* Vasospastic angina (positive test with acetylcholine),
* Evidence of cardiac ischemia,
* Coronary flow limiting myocardial bridge,
* Severe valvular disease
* Hospitalization for acute heart failure < 3 months
* Hypertrophic cardiomyopathy,
* Ejection fraction ≤ 30%,
* Permanent pacemaker or defibrillator leads in the right heart,
* Recent acute coronary syndrome < 6 months,
* Recent revascularization < 2 months,
* Right atrial pressure of 15 mmHg or higher,
* Severe renal impairment,
* Indication for cardiac resynchronization therapy,
* Pregnancy,
* Life expectancy of less than 1 year,
* Inclusion in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Clinical endpoint - Difference in summary Seattle Angina Questionnaire results between follow-up and baseline | 6 months
  The Seattle Angina Questionnaire (SAQ) is measured on a scale of 0 to 100 - higher scores represent better outcomes.
Mechanical endpoint - difference in left ventricle global longitudinal strain between follow-up and baseline | 6 months
  Left ventricle global longitudinal strain will be assessed with echocardiography. Measurements will be performed according to the current guidelines.

SECONDARY OUTCOMES:
Difference in Coronary Flow Reserve measured directly post-procedure and pre-procedure | Peri-procedural
Difference in Index of Microcirculatory Resistance and Resistance measured directly post-procedure and pre-procedure | Peri-procedural
Difference in Microvascular Resistance Reserve measured directly post-procedure and pre-procedure | Peri-procedural
  Microvascular Resistance Reserve will be assessed as the ratio of true resting to hyperemic microvascular resistance measured with thermodilution
Difference in Canadian Cardiovascular Society Class between follow-up and baseline | 6 months
  The Canadian Cardiovascular Society (CCS) classification ranges from Class I to IV - higher classes indicate more severe angina.
Difference in each Seattle Angina Questionnaire domain between follow-up and baseline | 6 months
  The Seattle Angina Questionnaire (SAQ) is measured on a scale of 0 to 100 - higher scores represent better outcomes.
Difference in Short Form-36 Health Survey results between follow-up and baseline | 6 months
  The Short Form-36 (SF-36) Health Survey is scored on a scale from 0 to 100 - higher scores indicate better health status and quality of life.
Difference in six-minute walk test between follow-up and baseline | 6 months
Difference in right ventricle four chamber longitudinal strain between follow-up and baseline | 6 months
Difference in left atrial strain conduit (%) between follow-up and baseline | 6 months
  Left atrial strain conduit (measured in %) will be assessed with echocardiography. Measurements will be performed according to the current guidelines.
Difference in left atrial strain pump (%) between follow-up and baseline | 6 months
  Left atrial strain pump (measured in %) will be assessed with echocardiography. Measurements will be performed according to the current guidelines.
Difference in left atrial strain reservoir (%) between follow-up and baseline | 6 months
  Left atrial strain pump (measured in %) will be assessed with echocardiography. Measurements will be performed according to the current guidelines.
Difference in average E/e' ratio between follow-up and baseline | 6 months
Difference in E (m/s) between follow-up and baseline | 6 months
  The parameter of mitral inflow (E - m/s) will be assessed with echocardiography. Measurements will be performed according to the current guidelines.
Difference in lateral, septal and average e' (cm/s) between follow-up and baseline | 6 months
  The e' (cm/s) will be assessed with echocardiography. Measurements will be performed according to the current guidelines.
Difference in Tricuspid Annular Plane Systolic Excursion between follow-up and baseline | 6 months
  Tricuspid Annular Plane Systolic Excursion (mm) will be assessed with echocardiography. Measurements will be performed according to the current guidelines.
Difference in RV S' (cm/s) between follow-up and baseline | 6 months
  RV S' (measured in cm/s) will be assessed with echocardiography. Measurements will be performed according to the current guidelines

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No